CLINICAL TRIAL: NCT05790096
Title: Phase 3 Randomized Clinical Effectiveness Study Clinical and Safety of Filgrastine® in Patients With Breast Cancer Treated With Myelotoxic Chemotherapy
Brief Title: Effectiveness and Safety Study of Filgrastine® in Patientes With Breast Cancer Treated With Myelotoxic Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Blau Farmaceutica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FILBLAU1022
Record Dates: First submitted 2023-01-13; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference Drug - Granulokine® (Active Comparator): Reference Drug - Granulokine® is presented in boxes containing vials containing 1,0 mL of solution for injection and 300µg of filgrastim.
  Granulokine® will be administered at a daily dose of 5 μg/kg of body weight, exclusively subcutaneously, according to randomization.
  Interventions: Biological: Granulokine
- Test Drug - Filgrastine® (Experimental): Test Drug -
  Filgrastine® is presented in boxes containing vials containing 1 mL of solution for injection and 300 µg of filgrastim.
  Filgrastine® will be administered at a daily dose of 5 μg/kg of body weight, exclusively subcutaneously, according to randomization.
  Interventions: Biological: Filgrastine

INTERVENTIONS:
Biological: Granulokine — Granulokine is presented in boxes containing vials containing 1,0 mL of solution for injection and 300µg of filgrastim.
  Arms: Reference Drug - Granulokine®
Biological: Filgrastine — Filgrastine is presented in boxes containing vials containing 1,0 mL of solution for injection and 300µg of filgrastim.
  Arms: Test Drug - Filgrastine®

SUMMARY:
Randomized Study of the Clinical Efficacy and Safety of Filgrastine® in Patients with Breast Cancer Treated with Myelotoxic Chemotherapy.

Primary Objective: to evaluate the activity and safety of Filgrastine® in Brazilian patients undergoing adjuvant treatment for breast cancer, with the frequency of grade 4 neutropenia in the first cycle of chemotherapy as the primary endpoint.

Secondary Objectives:

* Frequency of febrile neutropenia during treatment;
* Frequency of neutropenia of any degree in the first cycle;
* Frequency of hospitalization during treatment;
* Duration of grade 4 neutropenia in the first treatment cycle;
* Toxicity during treatment;
* Immunogenicity throughout treatment.

All endpoints will be descriptively analyzed in both groups of patients.

Study design Randomized (2:1), open-label, multicenter study.

Chemotherapy will be given on the first day of each cycle of treatment, for a maximum of four to eight cycles, depending on the regimen, patients whose chemotherapy treatment is prolonged beyond this period being withdrawn from the study.

Patients will be evaluated through laboratory tests, including complete blood count, biochemistry and anti-filgrastim antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Provision of the Free and Informed Consent Form by written;
* Female sex;
* Age between 18 and 75 years old;
* Diagnosis of breast cancer confirmed by cytology or histopathology;
* Disease in stages II or III, according to the classification tumor-node-metastasis (TNM);
* Indication of chemotherapy with full dose of one of the regimens eligible;
* Performance status of 0 or 1;
* Appropriate body functions (absolute neutrophil count [CAN] ≥1,500/mm³; platelet count ≥150,000/mm³; serum creatinine ≤1.2 mg/dL; bilirubin and transaminases ≤1.5 times the upper limit of normal).

Exclusion Criteria:

* Previous use of chemotherapy;
* Previous use of filgrastim;
* Prediction of prophylactic or therapeutic use of antibiotics, antifungals or antivirals in the first cycle of chemotherapy;
* Previous radiotherapy involving the pelvis or radiotherapy from any site within the last 6 weeks prior to randomization;
* History of bone marrow transplantation (as a recipient);
* Presence of other neoplasms;
* Presence of severe co-morbidities;
* Recent (<6 months) or planned participation in other studies clinical trials involving drugs of any nature or in studies of any form of intervention;
* Known intolerance or allergy to any of the components the filgrastim formulations evaluated in the study;
* Pregnancy or lactation (patients of childbearing potential must have a negative serological pregnancy test dated within 7 days prior to randomization).

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
frequency of grade 4 neutropenia in the first cycle of chemotherapy in the group of patients treated with Filgrastine® | 1 month

SECONDARY OUTCOMES:
Frequency of febrile neutropenia during treatment; | maximum 5 months
Frequency of neutropenia of any degree in the first cycle; | 1 month
Frequency of hospitalization during treatment; | maximum 5 months
Duration of grade 4 neutropenia in the first treatment cycle | 1 month
Adverse event monitoring | maximum 5 months
  Any adverse event that occurs from Treatment Visit 1 (first day of medication) onwards will be followed through to the Final Visit or until your resolution of the event, whichever is later
assessment of Immunogenicity throughout treatment by antigenic radiometric tests or ELISA | maximum 5 months
  The immunogenicity of filgrastim will be evaluated by antigenic radiometric tests or ELISA (enzyme-linked immunosorbant assay) to detect the formation of anti-G-CSF antibodies. All information will be recorded in the clinical form of the study.